CLINICAL TRIAL: NCT02689180
Title: Effect of Furosemide Withdraw in Stable Chronic Heart Failure Outpatients With Left Ventricular Dysfunction - the Brazilian Research Network on Heart Failure
Brief Title: Effect of Furosemide Withdraw in Stable Chronic Heart Failure Outpatients
Acronym: ReBIC-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-240
Record Dates: First submitted 2015-11-25; First posted 2016-02-23 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
Keywords: heart failure; diuretics; furosemide
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Withdraw of furosemide (Placebo Comparator): Withdraw of of 40 or 80 mg of furosemide per day
  Interventions: Drug: Placebo
- Maintenance of furosemide (Active Comparator): Maintenance of 40 or 80 mg of furosemide per day
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Placebo — Replacement of furosemide by placebo
  Arms: Withdraw of furosemide
Drug: Furosemide — Maintenance of furosemide on usual doses
  Arms: Maintenance of furosemide

SUMMARY:
The ReBIC-1 trial was designed to evaluate the potential clinical risks and benefits of withdrawing furosemide use in stable, apparently euvolemic, chronic HF outpatients in a multicentric double-blinded randomized clinical trial.

DETAILED DESCRIPTION:
Diuretics play a central role in HF treatment, particularly during episodes of acute decompensation. Furosemide is the prototype of loop diuretics, acting through the inhibition of the Na+K+2Cl- pump at the thick ascending limb of the Henle loop. According to international registries, almost all patients receive a loop diuretic during a hospital stay for acute decompensated HF and the majority are discharged taking a "maintenance dose". Despite the undeniable beneficial hemodynamic effects of improvement of peripheral and central congestion, the net clinical effect of the chronic use of diuretics on HF prognosis is controversial.

Observational studies suggest that use of high doses of diuretics might be related to unfavorable clinical consequences. Undesirable side effects of loop diuretics are not trivial and involve activation of the renin-angiotensin-aldosterone system, elevation of norepinephrine levels, increases in heart rate, detrimental effects on renal function and several electrolyte disturbances.

Few prospective clinical studies, however, directly evaluated the clinical risks and benefits of diuretics. Most of these studies were under-powered, performed more than 2 decades ago, before modern HF therapy with current drugs and devices was completely implemented.

Current clinical guidelines are unanimous to recommend use of diuretics in HF patients with clinical signs and symptoms of congestion, but reinforce the lack of solid clinical scientific evidence for its use, and the potential risks that might be involved. The European Society of Cardiology proposes the administration of the lowest dose necessary to achieve euvolemia, avoiding the unnecessary delay in the use of drugs that modify the natural history of the disease.

Based on these uncertainties about diuretic use in HF, the ReBIC-1 trial was designed to evaluate the potential clinical risks and benefits of withdrawing furosemide use in stable, apparently euvolemic, chronic HF outpatients in a multicentric double-blinded randomized clinical trial.

ReBIC is a Brazilian research network created to develop clinical studies in heart failure and composed predominantly by university tertiary care hospitals. ReBIC and the ReBIC-1 trial were sponsored by the Brazilian National Council for Scientific and Technological Development (CNPq, Brazil), a public governmental institution. Data collection, management, and analysis were performed at the network's data coordinating center at Hospital de Clínicas de Porto Alegre. All the authors reviewed and approved the manuscript and assume full responsibility for the accuracy and completeness of the data and for the fidelity of this report of the study protocol.

ReBIC-1 is a randomized, double-blind, parallel group, placebo-controlled, two-arm trial comparing the short-term efficacy and safety of discontinuation of furosemide in apparently euvolemic outpatients with chronic stable HF and reduced left ventricular ejection fraction (HF-REF).

ELIGIBILITY:
The ReBIC-1 study will enroll HF outpatients that fulfill the following criteria:

1. age equal or greater than 18 year-old;
2. New York Heart Association functional class I or II;
3. Left Ventricular Ejection Fraction ≤ 45% by transthoracic two-dimensional echocardiography performed within 3 months before the screening visit;
4. no previous HF related hospitalization or visit to emergency room within 6 months before the screening visit;
5. treatment with a stable dose of furosemide (40 or 80 mg per day) for at least 6 months before the screening visit;
6. plasma potassium < 5 mg/dl within 3 months before the screening visit;
7. optimal HF treatment with an angiotensin converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) and beta-blockers, unless contraindicated or not tolerated.

The ReBIC-1 study will exclude HF outpatients that fulfill the following criteria:

1. a clinical congestion score (CCS) > 5 points;
2. prior acute coronary syndrome, stroke or myocardial revascularization within 3 months before the screening visit;
3. any severe valve heart disease (aortic, mitral or tricuspid);
4. severe pulmonary disease (asthma, emphysema or fibrosis);
5. severe hepatic failure or cirrhosis;
6. end-stage acute or chronic renal disease (on hemodialysis);
7. malignancy on active treatment;
8. congenital heart disease;
9. participation on any other interventional clinical research;
10. inability to understand and sign informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility of furosemide withdraw - proportion of patients maintained without diuretic during follow-up | 90 days
  Proportion of patients maintained without diuretic during follow-up
Safety of furosemide withdraw - dyspnea score variation assessed by a visual analog scale | 90 days
  Dyspnea score variation assessed by a visual analog scale after randomization

SECONDARY OUTCOMES:
Variation of plasmatic levels of natriuretic peptides | Baseline and 90 days
  Levels of the N-terminal brain natriuretic peptide (NT pro-BNP)
Variation in meters walked assessed by the 6 minute walking test | Baseline and 90 days
Variation in renal function | Baseline, 15, 45 and 90 days
  Change in glomerular filtration rate ( ml/min /1.73 m²) estimated by the Modification of Diet in Renal Disease equation ( MDRD)
Variation on the Clinical Congestion Score | Baseline, 15, 45 and 90 days
  Clinical congestion score assessed by clinical history and physical examination (score from 1 to 22 point)
Clinical composite endpoints | 90 days
  Hospital admissions, emergency room visits and death within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Luis Eduardo Rohde, PHD, Study Chair — Hospital de Clínicas de Porto Alegre
Locations (1):
- Cardiovascular Division, Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lip GY, Gibbs CR, Beevers DG. ABC of heart failure: aetiology. BMJ. 2000 Jan 8;320(7227):104-7. doi: 10.1136/bmj.320.7227.104. No abstract available. PMID 10625270
- [Background] McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, Falk V, Filippatos G, Fonseca C, Gomez-Sanchez MA, Jaarsma T, Kober L, Lip GY, Maggioni AP, Parkhomenko A, Pieske BM, Popescu BA, Ronnevik PK, Rutten FH, Schwitter J, Seferovic P, Stepinska J, Trindade PT, Voors AA, Zannad F, Zeiher A; ESC Committee for Practice Guidelines. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012 Jul;33(14):1787-847. doi: 10.1093/eurheartj/ehs104. Epub 2012 May 19. No abstract available. PMID 22611136
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Cowley AJ, Stainer K, Wynne RD, Rowley JM, Hampton JR. Symptomatic assessment of patients with heart failure: double-blind comparison of increasing doses of diuretics and captopril in moderate heart failure. Lancet. 1986 Oct 4;2(8510):770-2. doi: 10.1016/s0140-6736(86)90298-9. PMID 2876233
- [Background] Eshaghian S, Horwich TB, Fonarow GC. Relation of loop diuretic dose to mortality in advanced heart failure. Am J Cardiol. 2006 Jun 15;97(12):1759-64. doi: 10.1016/j.amjcard.2005.12.072. Epub 2006 Apr 27. PMID 16765130
- [Background] Mielniczuk LM, Tsang SW, Desai AS, Nohria A, Lewis EF, Fang JC, Baughman KL, Stevenson LW, Givertz MM. The association between high-dose diuretics and clinical stability in ambulatory chronic heart failure patients. J Card Fail. 2008 Jun;14(5):388-93. doi: 10.1016/j.cardfail.2008.01.015. Epub 2008 May 27. PMID 18514930
- [Derived] Blacher M, Zimerman A, Engster PHB, Grespan E, Polanczyk CA, Rover MM, Neto JAF, Danzmann LC, Bertoldi EG, Simoes MV, Beck-da-Silva L, Biolo A, Rohde LE. Revisiting heart failure assessment based on objective measures in NYHA functional classes I and II. Heart. 2021 Sep;107(18):1487-1492. doi: 10.1136/heartjnl-2020-317984. Epub 2020 Dec 23. PMID 33361353
- [Derived] Rohde LE, Rover MM, Figueiredo Neto JA, Danzmann LC, Bertoldi EG, Simoes MV, Silvestre OM, Ribeiro ALP, Moura LZ, Beck-da-Silva L, Prado D, Sant'Anna RT, Bridi LH, Zimerman A, Raupp da Rosa P, Biolo A. Short-term diuretic withdrawal in stable outpatients with mild heart failure and no fluid retention receiving optimal therapy: a double-blind, multicentre, randomized trial. Eur Heart J. 2019 Nov 21;40(44):3605-3612. doi: 10.1093/eurheartj/ehz554. PMID 31424503